CLINICAL TRIAL: NCT01000961
Title: A Randomized, Crossover Pharmacokinetic and Pharmacodynamic Study to Determine the Safety and Efficacy of Cysteamine Bitartrate Delayed-release Capsules (RP103), Compared to Cystagon® in Patients With Nephropathic Cystinosis
Brief Title: Phase 3 Study of Cysteamine Bitartrate Delayed-release (RP103) Compared to Cystagon® in Patients With Cystinosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RP103-03
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Cystinosis
Keywords: cystinosis; cysteamine; inheritable disease; orphan disease; CTNS protein, human; metabolic disease; nephropathic cystinosis
MeSH Terms: conditions — Cystinosis; Rare Diseases; Metabolic Diseases | interventions — Cysteamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RP103 Q12H (Experimental)
  Interventions: Drug: Cysteamine Bitartrate Delayed-release Capsules (RP103)
- Cystagon® Q6H (Active Comparator)
  Interventions: Drug: Cystagon® (Cysteamine Bitartrate)

INTERVENTIONS:
Drug: Cystagon® (Cysteamine Bitartrate) — Run-in Period (Weeks 1, 2, 3) and Period 1 (Weeks 4, 5, 6) or Period 2 (Weeks 7, 8, 9); Immediate crossover to opposite treatment than taken during Period 1:
  Every 6H, supplied in 150 and 50mg capsules/Duration of Treatment: 3 weeks each period used
  Arms: Cystagon® Q6H
Drug: Cysteamine Bitartrate Delayed-release Capsules (RP103) — Period 1 (Weeks 4, 5, 6) or Period 2 (Weeks 7, 8, 9); Immediate crossover to opposite treatment than taken during Period 1:
  Every 12H, supplied in 75 and 25mg capsules/Duration of Treatment: 3 weeks
  Arms: RP103 Q12H

SUMMARY:
Cystinosis is an inherited disease that if untreated, results in kidney failure as early as the first decade of life. The current marketed therapy is Cystagon® (cysteamine bitartrate) which must be taken every six hours for the rest of the patient's life to prevent complications of cystinosis. RP103 is a formulation of cysteamine bitartrate that is being studied to see if it may be able to be given less frequently, once every 12 hours, and have similar results to four times a day Cystagon®.

DETAILED DESCRIPTION:
This is a multi-center, open-label, randomized, cross-over study to determine whether steady-state, twice a day treatment with Cysteamine Bitartrate Delayed-release Capsules(RP103) results in comparable depletion of white blood cell (WBC) cystine levels compared to the existing four times a day cysteamine treatment. It will involve up to 20 clinic visits plus intermittent home use of the RP103. Most of these clinic visits occur in clusters of 3-4 consecutive days. Eligible patients will be offered enrollment into a long-term follow up study.

Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects must have nephropathic cystinosis.
* Subjects must be on a stable dose of Cystagon® sufficient to maintain their white blood cell (WBC) cystine level at ≤ 1.0 nmol/half-cystine/mg protein.
* Subjects must be able to swallow their typically administered Cystagon® capsule with the capsule intact.
* Within the last 6 months, no clinically significant change in liver function [i.e., ALT, AST, total bilirubin] and renal function [i.e., estimated GFR] at Screening as determined by the Investigator.
* Subjects with an estimated GFR (corrected for body surface area) > 30 mL/min/1.73m2.
* Sexually active female subjects of childbearing potential (i.e., not surgically sterile [tubal ligation, hysterectomy, or bilateral oophorectomy] or at least 2 years naturally postmenopausal) must agree to utilize the same acceptable form of contraception from Screening through completion of the study.
* Subjects must be willing and able to comply with the study restrictions and requirements.
* Subjects or their or their parent or guardian must provide written informed consent and assent (where applicable) prior to participation in the study.

Exclusion Criteria:

* Subject's age < 6 years old or subject's weight < 21 kg.
* Subjects with a known history, currently of the following conditions or other health issues that make it, in the opinion of the investigator, unsafe for them to participate: inflammatory bowel disease (if currently active) or have had prior resection of small intestine; Heart disease (e.g., myocardial infarction, heart failure, arrhythmias or poorly controlled hypertension) 90 days prior to Screening; Active bleeding disorder 90 days prior to Screening; Malignant disease within the last 2 years.
* Patients with a hemoglobin level < 10 g/dL at Screening or a level that, in the opinion of the investigator, makes it unsafe for the subject to participate.
* Subjects receiving any form of cysteamine medication through a gastric tube.
* Subjects who are receiving maintenance dialysis or who have had a kidney transplant.
* Subjects who are on an active kidney transplant list or who are planning to receive a kidney transplant within 3 months of Screening.
* Subjects with known hypersensitivity to cysteamine or penicillamine.
* Female subjects who are nursing, planning a pregnancy, known or suspected to be pregnant, or have a positive serum pregnancy screen.
* Subjects who have a made a blood donation within 30 days of Screening.
* Subjects who, in the opinion of the Investigator, are not able or willing to comply with the protocol.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (8):
- United States (3):
  - Stanford University Medical School, Stanford, California
  - Emory Children's Center, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago (formerly Children's Memorial Hospital), Chicago, Illinois
- France (4):
  - Hospices Civils de Lyon, Lyon
  - Villeneuve-Lapeyronie Hospital, Montpellier
  - Necker Hospital, Paris
  - Robert Debre Hospital, Paris
- Radboud University Nijmegen Medical Center, Nijmegen, Netherlands

REFERENCES:
- [Background] Dohil R, Fidler M, Barshop BA, Gangoiti J, Deutsch R, Martin M, Schneider JA. Understanding intestinal cysteamine bitartrate absorption. J Pediatr. 2006 Jun;148(6):764-9. doi: 10.1016/j.jpeds.2006.01.050. PMID 16769383
- [Background] Fidler MC, Barshop BA, Gangoiti JA, Deutsch R, Martin M, Schneider JA, Dohil R. Pharmacokinetics of cysteamine bitartrate following gastrointestinal infusion. Br J Clin Pharmacol. 2007 Jan;63(1):36-40. doi: 10.1111/j.1365-2125.2006.02734.x. PMID 17229040
- [Background] Levtchenko EN, van Dael CM, de Graaf-Hess AC, Wilmer MJ, van den Heuvel LP, Monnens LA, Blom HJ. Strict cysteamine dose regimen is required to prevent nocturnal cystine accumulation in cystinosis. Pediatr Nephrol. 2006 Jan;21(1):110-3. doi: 10.1007/s00467-005-2052-0. Epub 2005 Oct 27. PMID 16252107
- See also: RP103 (marketed as PROCYSBI) is now approved by the US FDA for management of nephropathic cystinosis in patients 6 years and older — http://www.procysbi.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants randomized to each per sequence Arm are expected to remain in the same Arm throughout all intervention periods.
Groups:
- Cystagon First, Then Cystagon, Then RP103: Cystagon® dose in 50 mg and 150 mg capsule formulations administered every 6 hours in first intervention (after Run-in period) and RP103 dose in 25 mg and 75 mg capsule formulations administered every 12 hours in second intervention period.
- Cystagon First, Then RP103, Then Cystagon: RP103 dose in 25 mg and 75 mg capsule formulations administered every 12 hours in first intervention (after Run-in period) and Cystagon® dose in 50 mg and 150 mg capsule formulations administered every 6 hours in second intervention period.
Period: Run-in Period of 2-3 Weeks on Cystagon
Arm/Group | Cystagon First, Then Cystagon, Then RP103 | Cystagon First, Then RP103, Then Cystagon
Started | 21 (Part of the Safety analysis set) | 22 (Part of the Safety analysis set)
Completed | 21 | 22
Not Completed | 0 | 0
Period: First Intervention (3 Weeks)
Arm/Group | Cystagon First, Then Cystagon, Then RP103 | Cystagon First, Then RP103, Then Cystagon
Started | 21 | 22
Completed | 21 | 20
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Infection after pre-planned surgery | 0 | 1
Period: Second Intervention (3 Weeks)
Arm/Group | Cystagon First, Then Cystagon, Then RP103 | Cystagon First, Then RP103, Then Cystagon
Started | 21 | 20
Completed | 21 (Part of Efficacy analysis set) | 20 (Part of Efficacy analysis set)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were 39 participants analyzed for Cystagon®; and there were 37 participants analyzed for RP103.
Groups:
- RP103 and Cystagon® Crossover: Per Protocol Population
Arm/Group | RP103 and Cystagon® Crossover
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.9 (4.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 23
Region of Enrollment [Number; unit: participants]
  France | 13
  United States | 22
  Netherlands | 4

OUTCOME MEASURES:

1. Primary Outcome: The Steady-state White Blood Cell Cystine Levels of RP103 Compared to Cystagon®
Time Frame: 4 weeks after the last subject has completed the study
Measure: Least Squares Mean (Standard Error); unit: nmol ½ Cystine / mg protein
Groups:
- RP103; Cystagon®: Per Protocol Population
Arm/Group | RP103 | Cystagon®
Number analyzed (Participants) | 39 | 39
nmol ½ Cystine / mg protein | 0.5152 (0.05555) | 0.4367 (0.05555)
Statistical Analysis 1: Comparison: RP103 vs Cystagon®; 16-subject study will have 90% power to reject the null hypothesis of non-inferiority at the 0.025 level of significance with a non-inferiority margin of 0.3. Final analysis was performed at a nominal significance level of 0.02104; Test type: Non-Inferiority or Equivalence — The non-inferiority endpoint of the clinical trial would be achieved if the upper limit of the 95.8% CI of the difference between RP103 and Cystagon® was less than the a-priori 0.3 non-inferiority margin, which would correspond to an observed p-value less than or equal to 0.02104; p = 0.0001, t-test, 1 sided; Mean Difference (Final Values) = 0.0785, 95.8% CI 2-sided [0.0107 to 0.1464] — 95.8% confidence interval was used instead of 95% to take into account a sample size re-estimation calculation that was performed after 20 patients were enrolled

2. Secondary Outcome: Comparison of Cysteamine PK Profiles, Steady State Cmax, Between RP103 and Cystagon®.
Time Frame: 4 weeks after the last subject has completed the study
Measure: Least Squares Mean (Standard Deviation); unit: Cmax (mg/L)
Arm/Group | Cystagon® | RP103
Number analyzed (Participants) | 39 | 37
Cmax (mg/L) | 2.73 (1.36) | 3.70 (1.72)
Statistical Analysis 1: Comparison: Cystagon® vs RP103; Test type: Superiority or Other; Median Difference (Final Values) = 1.40, 95% CI 2-sided [1.17 to 1.67]

3. Secondary Outcome: Comparison of Cysteamine PK Profiles, Steady State Tmax, Between RP103 and Cystagon®.
Time Frame: 4 weeks after the last subject has completed the study
Measure: Least Squares Mean (Standard Deviation); unit: Tmax (minute)
Arm/Group | Cystagon® | RP103
Number analyzed (Participants) | 39 | 37
Tmax (minute) | 72 (31) | 187 (89)
Statistical Analysis 1: Comparison: Cystagon® vs RP103; Test type: Superiority or Other; Mean Difference (Final Values) = 105, 95% CI 2-sided [90 to 150]

4. Secondary Outcome: Comparison of Cysteamine PK Profiles, AUC(0-t), Between RP103 and Cystagon®.
Time Frame: 6 hours post dosing for Cystagon®; 12 hours post dosing for RP103.
Measure: Least Squares Mean (Standard Deviation); unit: AUC(0-t) (min*mg/L)
Arm/Group | Cystagon® | RP103
Number analyzed (Participants) | 39 | 37
AUC(0-t) (min*mg/L) | 357 (150) | 739 (334)
Statistical Analysis 1: Comparison: Cystagon® vs RP103; Test type: Superiority or Other; Mean Difference (Final Values) = 2.03, 95% CI 2-sided [1.75 to 2.39]

ADVERSE EVENTS:
Time Frame: Treatment periods
Description: Safety population AE reporting
Groups:
- RP103; Cystagon®: Safety Population during treatment periods
Arm/Group | RP103 | Cystagon®
Serious Adverse Events (participants affected / at risk) | 6/43 | 1/41
Other Adverse Events (participants affected / at risk) | 16/43 | 5/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RP103 (N=43) | Cystagon® (N=41)
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RP103 (N=43) | Cystagon® (N=41)
Vomiting (Gastrointestinal disorders) | 5 (8) | 3 (5)
Nausea (Gastrointestinal disorders) | 5 (7) | 2 (3)
Abdominal Pain (Gastrointestinal disorders) | 3 (4) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators may publish or disclose study data, with the restriction that sponsor may embargo such communications for a period up to 60 days from the time submitted to sponsor. As a multi-center study, first publication of results will take place in conjunction with all investigators. If such a multi-center publication is not forthcoming within 18 months of study completion, individual investigators may publish as restricted according to limitations expressed above (60 day embargo).